CLINICAL TRIAL: NCT07131774
Title: Evaluation of a Diary for Assessing Treatment Outcomes in Patients With Pulmonary Infections Caused by Nontuberculous Mycobacteria (NTM)
Brief Title: Treatment Monitoring for NTM Infections With a Symptom Diary
Acronym: NTMdiary
Status: Recruiting | Type: Observational
Sponsor: Research Center Borstel (Other)
Responsible Party: Principal Investigator, Thomas Theo Brehm, Dr. med., Research Center Borstel
Other Study IDs: NTMdiary2025-002
Record Dates: First submitted 2025-04-29; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Non-Tuberculous Mycobacterial (NTM) Infections
Keywords: symptom diary; microbiology; radiology
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NTM infection, under therapy: Patients who have a pulmonary NTM infection according to ATS/IDSA criteria and are receiving antimicrobial therapy (Cohort 1).
  Interventions: Other: Filling in a symptom diary
- NTM infection, no therapy: Patients who have a pulmonary NTM infection according to ATS/IDSA criteria but are not receiving therapy due to a clinical decision or the patient's own choice (Cohort 2).
  Interventions: Other: Filling in a symptom diary

INTERVENTIONS:
Other: Filling in a symptom diary — Each patient will receive a diary form in which they are asked to record their symptoms, body temperature, and body weight on a daily basis. This approach is intended to provide a comprehensive overview of the disease course and the impact of treatment over time.
  Depending on hospitalization status, disease severity, treatment progress, and national treatment guidelines, clinical, microbiological, and radiological follow-up assessments will be performed as part of routine care at intervals ranging from weekly to monthly. No additional study visits or microbiological or radiological diagnostics outside of standard clinical care will be conducted.

SUMMARY:
The primary aim of the study is to investigate the correlation between patient-reported symptoms recorded in the diary and the microbiological and radiological disease course in patients with pulmonary infections caused by nontuberculous mycobacteria (NTM).

DETAILED DESCRIPTION:
This prospective observational study investigates the suitability of a symptom diary for assessing disease progression and treatment outcomes in patients with pulmonary infections caused by nontuberculous mycobacteria (NTM). The aim of the study is to correlate the symptoms documented in the diary with microbiological and radiological parameters to gain a better understanding of the disease course and treatment effects. This may contribute to the development of a simpler and non-invasive tool that could improve patients' quality of life and enable more precise monitoring of disease progression.

This multicenter study plans to enroll 200 adult patients with confirmed pulmonary NTM infections who are capable of providing informed consent. Each patient will document daily symptoms - such as cough, body weight, temperature, and other complaints - in a symptom diary over a period of six months. In addition, clinical routine data, including microbiological and radiological findings, will be used without requiring any additional diagnostic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary NTM infection according to ATS/IDSA criteria (1)
* Age ≥ 18 years
* Ability to provide informed consent
* Willingness to participate in the study AND
* Clinical decision to initiate antimicrobial therapy as part of routine care

  * Cohort 1 OR
* Clinical decision against antimicrobial therapy as part of routine care

  * Cohort 2

Exclusion Criteria:

* Lack of ability to provide informed consent
* Language barriers that prevent completion of the diary
* Antimicrobial therapy for the NTM infection already initiated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 18 years of age, including women of childbearing potential with or without contraception. Only adult patients capable of giving informed consent will be included; obtaining consent from legal guardians is not planned.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Degree of correlation of the symptom diary with radiology | 6 months from enrolement
  The primary endpoint of the study is the degree of correlation between patient-reported symptoms recorded in the diary in patients with pulmonary infections caused by nontuberculous mycobacteria (NTM) and the radiological course of the disease.
  Radiological course of the disease is assessed by a radiological composit measure consisting of an ordinal scale for nodule extent, consolidation extent, bronchiectasis severity and -extent, mucus plugging, cellular bronchiolitis severity and -extent, cavity diameter, -wall thickness, and number of cavities. Worsening (+1, step up) and improvement (-1 step down) are added and show overall worsening (>= +1), overall improvement (<= -1) or stable disease (= +/-0).
Degree of correlation of the symptom diary with microbiology | 6 months from enrolment
  The primary endpoint of the study is the degree of correlation between patient-reported symptoms recorded in the diary in patients with pulmonary infections caused by nontuberculous mycobacteria (NTM) and the microbiological course of the disease, assessed by
  - the mycobacterial load in sputum microscopy
Degree of correlation of the symptom diary with microbiology | 6 months from enrolment
  The primary endpoint of the study is the degree of correlation between patient-reported symptoms recorded in the diary in patients with pulmonary infections caused by nontuberculous mycobacteria (NTM) and the microbiological course of the disease, assessed by
  - time to positivity in liquid culture
Degree of correlation of the symptom diary with microbiology | 6 months from enrolment
  The primary endpoint of the study is the degree of correlation between patient-reported symptoms recorded in the diary in patients with pulmonary infections caused by nontuberculous mycobacteria (NTM) and the microbiological course of the disease, assessed by
  - treatment duration until culture conversion (defined as the absence of detectable mycobacteria using the aforementioned methods)

SECONDARY OUTCOMES:
Degree of correlation between the symptom diary and further treatment monitoring parameters | 6 months from enrolement
  Degree of correlation between patient-reported symptoms recorded in the diary and the radiological course of disease in patients with pulmonary infections caused by nontuberculous mycobacteria.
  Radiological course of the disease is assessed by a radiological composit measure consisting of an ordinal scale for nodule extent, consolidation extent, bronchiectasis severity and -extent, mucus plugging, cellular bronchiolitis severity and -extent, cavity diameter, -wall thickness, and number of cavities. Worsening (+1, step up) and improvement (-1 step down) are added and show overall worsening (>= +1), overall improvement (<= -1) or stable disease (= +/-0).
Degree of correlation between the symptom diary and further treatment monitoring parameters | 6 months from enrolement
  Differences in the severity and development of symptoms during the course of treatment depending on the mycobacterial subspecies.
Degree of correlation between the symptom diary and further treatment monitoring parameters | 6 months from enrolement
  Degree of correlation between patient-reported symptoms recorded in the diary over the course of the study and the use of antimicrobial therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Lange, Prof. Dr. med. Dr. h.c., Study Chair — Clinical Infectious Diseases, Research Center Borstel, Leibniz Lung Center
Locations (3):
- Germany (3):
  - Abteilung Infektiologie, Klinik für Innere Medizin II, Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Schwerpunkt Infektiologie, Medizinische Klinik 2, Zentrum für Innere Medizin, Universitätsmedizin Frankfurt, Frankfurt am Main, Hesse
  - Pulmonary Care Center, Research Center Borstel, Leibniz Lung Center, Borstel, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request.
Supporting Information: Study Protocol, ICF